CLINICAL TRIAL: NCT01585610
Title: Motivating Smokers With Mobility Impairments to Quit Smoking
Acronym: ABLE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Belinda Borrelli, Professor of Psychiatry and Human Behavior, Brown University School of Medicine, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01CA137616-01 (NIH)
Record Dates: First submitted 2012-04-20; First posted 2012-04-26 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Smoking
Keywords: smoking; smoking cessation; disabled persons; behavioral research
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DVD Program (Experimental)
  Interventions: Behavioral: DVD Intervention
- Standard Care Printed Materials (Active Comparator)
  Interventions: Behavioral: Standard Care Printed Materials

INTERVENTIONS:
Behavioral: DVD Intervention — Four theory-based intervention DVDs will be provided to participants in this arm, the first in the home after Baseline assessment and the next 3 at 1-month intervals by mail. DVDs focus on motivating smoking cessation among people with mobility impairments using Behavioral Activation as the primary theoretical construct. Short (< 5 min.) phone calls will also be placed to each participant in between DVD deliveries and after receipt of DVD 4.
  Other Names: Behavioral Activation; Video; Home Intervention; People with Disabilities; Smoking Cessation
  Arms: DVD Program
Behavioral: Standard Care Printed Materials — Four sets of standard smoking cessation printed materials will be provided to participants in this arm, the first in the home after Baseline assessment and the next 3 at 1-month intervals by mail. Short (< 5 min.) phone calls will also be placed to each participant in between materials deliveries and after the 4th and final set is sent by mail.
  Other Names: Print Materials; Home Intervention; People with Disabilities; Smoking Cessation
  Arms: Standard Care Printed Materials

SUMMARY:
The purpose of this study is to determine if a newly designed DVD program performs better than standard, printed quit-smoking materials to help smokers who have mobility limitations (e.g., use a cane, wheelchair, braces, crutches, prosthesis) to quit smoking.

DETAILED DESCRIPTION:
People with physical disabilities (mobility impairments) who use assistance to ambulate have higher smoking rates (32.5%) when compared to people who have a disability and do not need assistance (23%) and when compared to people who are not disabled (19.8%; Brawarsky et al. 2002). The aims of the current study are to: 1) develop a series of theory-based Intervention DVDs focused on motivating smoking cessation among people with mobility impairments (i.e., chronically use some type of assistance to walk such as walker, cane, wheelchair, braces, etc) and 2) test the efficacy of the Intervention DVDs versus Print-Based Standard Care among 560 smokers with mobility impairments in a randomized trial. The materials in both groups will be mailed on a monthly basis for four months, and are organized in separate sections according to readiness to quit. Participants in both groups will receive a) nicotine patches at no cost if they are ready to quit and b) brief phone calls (~5 minutes) between mailings to assess and encourage viewing the materials. We hypothesize that smokers who are randomized to receive the Intervention DVDs will be significantly more likely to achieve 7-day and 30-day point-prevalence abstinence at 1 and 6 month follow-ups vs. those who receive Print-Based Standard Care. The Intervention DVDs will be based on Behavioral Activation Theory, and address specific barriers to quitting in this population (increased stress, decreased positive affect, increased depressed mood, activity restriction, and self-efficacy). We hypothesize that the intervention will impact these mediators directly, as well as indirectly through Behavioral Activation (goal setting and pleasant activities). If effective, our DVD intervention could have a high level of public health and clinical significance, as it could be easily disseminated at low cost through national disability-related organizations, networks of independent living centers, or physician offices. It will also substantially improve the health and quality of life for people with physical disabilities.

ELIGIBILITY:
Inclusion Criteria:

* chronic use of some type of assistance to walk (e.g., walker, cane, wheelchair, braces)

  * at least one year duration of the physical disability
* ability to speak and understand English
* smoke > 3 cigarettes per day and > 100 cigarettes in their lifetime

  * 18 years of age or older
  * visual capability to the extent that they can view the video and potentially benefit from it.

Exclusion Criteria:

* current receipt of hospice care
* temporary mobility impairment
* refusal to be tape-recorded
* pregnant or lactating
* severe cognitive impairments that would significantly compromise their ability to complete questionnaires or participate in the intervention (a Telephone Interview of Cognitive Status Mini-Mental State score < 25)
* current severe psychiatric or substance abuse problems (> 14 alcoholic drinks per week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-08 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Smoking Status: 7-day and 30-day point prevalence | 1 and 6 months Post-Intervention
  Seven-day point prevalence abstinence (no smoking at all in the previous seven days) will be assessed by self-report. We will also assess 30 day point-prevalence abstinence (no smoking at all in the previous 30 days) by self-report. Participants who have switched to other forms of tobacco will be considered "smokers." Participants who self-report no smoking will be asked to provide a Carbon Monoxide (CO) breath sample. Participants who have a CO < 10ppm will be considered abstinent.

SECONDARY OUTCOMES:
Participant Satisfaction | 2, 6, 10, and 14 weeks after Baseline
  Participant satisfaction will be assessed during phone calls in the intervention period in two ways: 1) the Educational Materials Review Form Questionnaire (EMRFQ), and 2) participants' open-ended opinions about the most recent mailing (what they liked most, least, did they retain the video/print-based material, and was there anything objectionable). These will be used to evaluate DVDs and print material on: ease of use and understanding, degree of helpfulness, ability to attract attention and change behavior, and usefulness for national distribution.
Use of Intervention Materials | 2, 6, 10, and 14 weeks after Baseline
  During follow-up phone calls in between mailings we will assess the length of time spent watching the video or reading the print materials, segments viewed or chapters read, and whether others in the household viewed the video or print-based materials. Participants will be asked simple recall questions about segments viewed or chapters read (characters, storyline, etc.) so that those who viewed the materials will be able to answer them easily.
Motivation to Quit | Baseline & 1 and 6 mos Post-Intervention
  We will use the Contemplation Ladder.205 Validity studies have shown associations with cognitive and behavioral indices of readiness to consider smoking cessation and with making quit attempts (e.g., intention to quit, nicotine dependence).We will also assess Stage of Change to compare its predictive and concurrent validity with this measure. We will assess motivation at baseline to assess equivalency between groups, and analyze as a covariate if necessary.
Self-Efficacy | Baseline & 1 and 6 mos Post-Intervention
  The Generalized Self-Efficacy Scale is a 10-item scale that assesses one's belief in the ability to respond and cope with novel or difficult situations and unexpected setbacks or obstacles. Self-efficacy to quit smoking will be assessed with a 15-item version of the Confidence Questionnaire. We will assess the mediational role of both general and specific self-efficacy in predicting outcome.
Depressed Mood | Baseline & 1 and 6 mos Post-Intervention
  Depressed Mood will be assessed with the 20-item Center for Epidemiologic Studies Depression Scale (CES-D210). Depressed mood is associated with difficulty quitting smoking and staying quit.Our DVD intervention will target depressed mood and assess a mediator of treatment outcome.
Perceived Stress | Baseline & 1 and 6 mos Post-Intervention
  The 4-item Perceived Stress Scale will be used to assess the degree to which participants perceive their environment and their experiences as stressful. The scale correlates well with scores on life-event measures, and has demonstrated good reliability. Our intervention will target stress because levels of stress can impact quitting and because a number of studies have found that persons with physical disabilities report elevated perceived stress scores. Our DVD Intervention will target stress and assess its role as a mediator of treatment outcome
Positive Affect | Baseline & 1 and 6 mos Post-Intervention
  We will use the Positive and Negative Affect Scale (PANAS; Watson et al 1998). The PANAS is a self-report state mood questionnaire that has a positive and negative affect subscale. Positive affect has been associated with quitting smoking and is a predictor of health and disability across many samples. Our DVD Intervention will target positive affect and we will assess the role of positive affect as a mediator of treatment outcome.
Behavioral Activation: Goal Setting and Achievement | Baseline & 1 and 6 mos Post-Intervention
  (Borrelli & Mermelstein). Subgoal setting will be the total number of goals set since last contact. Subgoal achievement will be the number of goals met between assessments vs the number of goals set for that time period. We will examine whether number of goals set, proportion of goals achieved, or the type of subgoal achieved (direct or indirect), have effects on follow-up smoking status. We will assess this measure as a mediator of treatment outcome.
Behavioral Activation: Pleasant activities | Baseline & 1 and 6 mos Post-Intervention
  The Pleasant Events Schedule measures an individual's frequency and subjective pleasure of various potentially reinforcing events and activities. Activities cover two primary areas: passive or active and social or non-social. Participants rate each item for frequency during the past month, and subjective enjoyability during that same month. We will assess this measure as a mediator of treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Borrelli, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Busch AM, Borrelli B. Valued life activities and readiness to quit smoking among mobility-impaired smokers. Health Psychol. 2012 Jan;31(1):122-5. doi: 10.1037/a0025218. Epub 2011 Aug 29. PMID 21875204